CLINICAL TRIAL: NCT01876238
Title: Feasibility of a Team Approach for Discussing Prognosis and Treatment Goals With Patients Diagnosed With Advanced Breast Cancer
Brief Title: Feasibility of a Team Approach for Discussing Prognosis and Treatment Goals in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE12112
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Advanced Breast Cancer; Stage 4 Breast Cancer; Recurrent Breast Cancer
Keywords: Breast Cancer; Patient-Doctor Communication; Supportive Care
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- T-PAT Intervention (Experimental): Prognosis discussion intervention with study team.
  Interventions: Other: T-PAT; Other: Surveys
- Control: Standard Care (Active Comparator): Usual care appointment
  Interventions: Other: Surveys

INTERVENTIONS:
Other: T-PAT
  Arms: T-PAT Intervention
Other: Surveys — Pre-test and posttest surveys and questionnaires
  Other Names: State Hope Scale; Tolerate Adverse States Survey; Physical Functioning Measure (MOS-PF); Beleif in CUrability (BIC); Illness Uncertainty Survey; Treatment Goal Preference Questionnaire

SUMMARY:
This research study will examine how patients with advanced breast cancer and their oncology team communicate and plan ongoing care.The purpose of this study is to find out more about care planning during advanced breast cancer. The study will see if certain aspects of communication make a difference in how patients understand their illness.

DETAILED DESCRIPTION:
The new communication practice (T-PAT) is a team approach for discussing prognosis and treatment goals. T-PAT is specifically designed to a) increase understanding of the prognosis and treatment goal, b) decrease illness uncertainty, and c) help the patient preserve hope for the future.This dedicated clinical visit features a structured discussion of prognosis, treatment goals and options, and end of life concerns. The planned team discussion will include information contributions for the treating medical oncologist, an oncology nurse and social worker who currently work together to provide breast cancer care.

Primary Objectives:

1. Assess the feasibility of implementing the T-PAT prognosis discussion intervention.
2. Compare the effects of T-PAT vs. usual care on pertinent patient reported outcomes including: a) understanding of the prognosis and treatment goal, b) illness uncertainty, and c) hope.

   * First, a survey will be administered to patients in the waiting room before the next office visit. This should take 15-20 minutes.
   * The second part involves participating in a scheduled appointment that will be audio-recorded and focus on sharing information about the patient's illness. Patients will be randomized to either participate in an appointment featuring new communication practices (T-PAT)or a regular care appointment.
   * The third part involves a 20 minute survey, after the appointment, with a member of the study staff. This will take place over the telephone one or two days after the appointment.
   * The fourth part is completion of a written reflection on the patients participation in the study, which will be returned in a pre-addressed, stamped envelope. Generally, this should take about 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Women newly or currently diagnosed with stage 4 or recurrent breast cancer
* Patients of Dr. Paula Silverman at Seidman Cancer Center
* Ambulatory
* Able to understand and participate in a discussion about their disease progression

Exclusion Criteria:

* Hospitalized
* Unable to speak English
* Unable to attend an office visit
* ECOG performance score of >3

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of Implementing the T-PAT Prognosis Discussion Intervention | 8 months
  Accuracy and completion rate of the planned intervention components will be observed.

SECONDARY OUTCOMES:
Patient Recorded Measures: Hope | 8 months
  Using the Snyder et al.'s State Hope Scale
Patient Recorded Measures: Willingness to Tolerate Adverse States | 8 months
  Six-Item scale that measures motivation to endure burden associated with aggressive care. Higher scores indicate a greater willingness to tolerate adverse states.
Patient Recorded Measures: Medical Outcomes Study-Physical Functioning Measure (MOS-PF) | 8 months
  Assess patient physical function
Patient Recorded Measures: Belief in Curability (BIC) | 8 months
  Assess patients perceptions about prognosis independent of what they recall being told by their doctor.
Patient Recorded Measures: Illness Uncertainty | 8 months
  16-item scale tapping patient uncertainty about symptoms, diagnosis, treatment, and future plans.
Patient Recorded Measures: Treatment Goal Preference | 8 months
  Patients will be asked to report their preference for aggressive care.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Step, PhD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States